CLINICAL TRIAL: NCT00047294
Title: Phase II Study Of Temozolomide, Thalidomide And Celecoxib In Patients With Newly Diagnosed Glioblastoma Multiforme In The Post-Radiation Setting
Brief Title: Temozolomide, Thalidomide, and Celecoxib Following Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Patrick Y. Wen, MD, Director, Center for Neuro-Oncology, Dana-Farber Cancer Institute
Masking: None | Purpose: Treatment
Other Study IDs: 00302; P30CA006516 (NIH); CDR0000257587; NCI-G02-2118; CELGENE-2000-P-002521/1
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2005-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult mixed glioma; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioma; Glioblastoma; Gliosarcoma | interventions — Celecoxib; Temozolomide; Thalidomide; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: celecoxib
Drug: temozolomide
Drug: thalidomide
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide and celecoxib may stop the growth of tumor cells by stopping blood flow to the tumor and may increase the effectiveness of temozolomide by making tumor cells more sensitive to the drug.

PURPOSE: Phase II trial to study the effectiveness of combining temozolomide, thalidomide, and celecoxib following radiation therapy in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of adjuvant temozolomide, thalidomide, and celecoxib after radiotherapy, in terms of time to tumor progression and overall survival, in patients with newly diagnosed glioblastoma multiforme.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral temozolomide once daily on days 1-5 and oral thalidomide once daily and oral celecoxib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial glioblastoma multiforme or gliosarcoma
* Completed standard external beam radiotherapy within the past 5 weeks
* Stable disease by MRI or CT scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 4 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* No history of bleeding disorder

Hepatic

* Bilirubin less than 1.5 mg/dL
* SGPT less than 2.5 times normal
* Alkaline phosphatase less than 2.5 times normal

Renal

* BUN less than 1.5 times upper limit of normal (ULN) OR
* Creatinine less than 1.5 times ULN

Cardiovascular

* No deep vein thrombosis within the past 3 weeks (must be clinically stable)

Pulmonary

* No pulmonary embolism within the past 3 weeks (must be clinically stable)

Other

* Must participate in System for Thalidomide Education and Prescribing Safety program
* No peripheral neuropathy grade 2 or greater
* No active infection
* No concurrent illness that may obscure toxicity or dangerously alter drug metabolism
* No other serious concurrent illness
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception for 1 month before, during, and for 1 month after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior thalidomide
* No concurrent immunotherapy
* No concurrent prophylactic filgrastim (G-CSF)

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy
* Concurrent corticosteroids must be at stable or decreasing dose over the past 7 days

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* No concurrent surgery

Other

* No other concurrent anticancer therapy
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y. Wen, MD, Study Chair — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Center at the University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Result] Kesari S, Schiff D, Henson JW, Muzikansky A, Gigas DC, Doherty L, Batchelor TT, Longtine JA, Ligon KL, Weaver S, Laforme A, Ramakrishna N, Black PM, Drappatz J, Ciampa A, Folkman J, Kieran M, Wen PY. Phase II study of temozolomide, thalidomide, and celecoxib for newly diagnosed glioblastoma in adults. Neuro Oncol. 2008 Jun;10(3):300-8. doi: 10.1215/15228517-2008-005. Epub 2008 Apr 10. PMID 18403492